CLINICAL TRIAL: NCT06303310
Title: Comparative Effects of Gaze Stability Exercises and Optokinetic Exercises on Dizziness, Balance and Activities of Daily Living in Patients With Vestibular Hypofunction
Brief Title: Comparative Effects Of Gaze Stability Exercises And Optokinetic Exercises In Patients With Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0296
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Vestibular Disorder
Keywords: Optokinetic exercises, Vestibular hypofunction,
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Group A (Gaze Stability Exercises + Balance Exercises) Group B (Optokinetic Exercises + Balance Exercises)
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blinded. Assessor will be the person having 10 years experience in neuromuscular rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive gaze stability exercises consist of 5 structured components for 20 minutes and the routine physical therapy consisting of balance exercises of 20 minute for 5 days a week for 4 weeks.
  Interventions: Other: Gaze Stability Exercises; Other: Routine Physical Therapy
- Group B (Experimental): Group B will receive optokinetic exercises for 20 minutes and the routine physical therapy consisting of balance exercises of 20 minute for 5 days a week for 4 weeks.
  Interventions: Other: Optokinetic Exercises; Other: Routine Physical Therapy

INTERVENTIONS:
Other: Gaze Stability Exercises — Group A ( Gaze Stability Exercise+ Routine Physical Therapy) Group A will receive gaze stability exercises consist of 5 structured components for 20 minutes and the routine physical therapy consisting of balance exercises of 20 minute for 5 days a week for 4 weeks.(16)
  Other Names: Optokinetic Exercises
  Arms: Group A
Other: Optokinetic Exercises — Group B (Optokinetic Exercises+Routine Physical Therapy) Group B will receive optokinetic exercises for 20 minutes and the routine physical therapy consisting of balance exercises of 20 minute for 5 days a week for 4 weeks
  Arms: Group B
Other: Routine Physical Therapy — Routine Physical Therapy

SUMMARY:
This randomized clinical trial will occur at Bahawal Victoria Hospital, Bahawalpur within 7 months after the approval of synopsis. The sample size for this trial will be 40 participants. Participants fulfilling the inclusion criteria will be recruited by using the convenience sampling randomly allocated into two groups by computer generator method. 20 participants will be assigned to Group A receiving gaze stability exercises and 20 to the Group B receiving optokinetic exercises, both alongside routine physical therapy. Each group will undergo 5 weekly sessions of treatment for 4 weeks.The assessment tools include Dizziness Handicap Inventory for dizziness; Mini-BESTest and modified-Clinical Test of Sensory Interaction of Balance for balance assessment while Vestibular Disorders Activities of Daily Living Scale for daily activities.

DETAILED DESCRIPTION:
Vestibular hypofunction characterized by impaired balance and spatial orientation due to the inner ear's vestibular system issues present significant challenges for affected individuals. Gaze stability exercises enhance focus despite head movements while optokinetic exercises improve eye movement control. Both interventions benefit people with vestibular issues aiming to enhance stability, decrease dizziness and improve balance. This study aims to investigate and compare the effects of gaze stability exercises and optokinetic exercises on dizziness, balance, and activities of daily living in patients with vestibular hypofunction.

This randomized clinical trial will occur at Bahawal Victoria Hospital, Bahawalpur within 7 months after the approval of synopsis. The sample size for this trial will be 40 participants. Participants fulfilling the inclusion criteria will be recruited by using the convenience sampling randomly allocated into two groups by computer generator method. 20 participants will be assigned to Group A receiving gaze stability exercises and 20 to the Group B receiving optokinetic exercises, both alongside routine physical therapy. Each group will undergo 5 weekly sessions of treatment for 4 weeks.

The assessment tools include Dizziness Handicap Inventory for dizziness; Mini-BESTest and modified-Clinical Test of Sensory Interaction of Balance for balance assessment while Vestibular Disorders Activities of Daily Living Scale for daily activities. Assessment will be carried out at baseline, 2nd and 4th week. The data will be analyzed using SPSS version 24 for Windows software with the significance level set at p = 0.05. Shapiro-Wilk test will assess data normality. Between group analysis will utilize the Independent t-test for parametric data and Mann-Whitney test for non-parametric data. Within group comparisons will employ repeated measure ANOVA Paired t- test for parametric data and Friedman ANOVA for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

Participants will be of both genders. Participants age will be between 23 to 63 years. Participants diagnosed with unilateral vestibular disorders by ENT specialist. Individuals who have MOCA score ≤26. Participants with positive head thrust test. Participants with positive supine roll test.

Participants have one or more of the following characteristics:

Related burden symptoms that affected their daily activities. A history of dizziness/vertigo triggered by head or body movement.

Exclusion Criteria:

Individuals with a history of neurological or psychological deficit. Individuals with the diagnosis of benign paroxysmal positional vertigo as individuals.

Individuals who had a previous surgery that could affect balance or cause dizziness.

Individuals with orthopedic problems that prohibited the performance of the exercise and that impact one's balance and walking pattern.

Individuals who report spontaneous episodes of dizziness, which are not worsened by movements Individuals which are completely dependent on the assistive device during mobility.

Imbalance due to diabetic neuropathy.

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | At Baseline, 2nd week and 4th week
  The Dizziness Handicap Inventory sees widespread use in evaluating disability associated with dizziness.The DHI comprises 25 questions, with seven pertaining to physical aspects, nine to the emotional domain, and nine to functional aspects.
Mini-Bestest | At Baseline, 2nd week and 4th week.
  Mini Balance Evaluation Systems Test is used to evaluate the balance performance. It consists of 14 tasks, each scored on a three-level scale: 0 for severe inability to perform, 1 for moderate performance, and 2 for normal performance, resulting in a total possible score of 28.
Modified-Clinical Test of Sensory Interaction on Balance | At Baseline, 2nd week and 4th week.
  The Clinical Test of Sensory Interaction on Balance was specifically designed to evaluate how the visual, somatosensory, and vestibular systems contribute to postural control.Individuals experiencing uncompensated peripheral vestibular loss might encounter challenges in maintaining an upright posture, particularly when there are alterations in visual input and support surface conditions. Prior to the test, patients are positioned on the platform designated for the evaluation. Throughout each phase of the assessment, patients are instructed to stand steadily and sustain their position on the platform for 30 seconds. The duration of time the patients remained standing is documented during each trial, repeated three times in total, and an average is calculated based on these three trials
Vestibular Disorders Activities of Daily Living Scale | At Baseline, 2nd week and 4th week.
  The Vestibular Disorders Activities of Daily Living Scale holds significant importance as it focuses on examining daily activities that may be adversely affected by vestibular disorders.Comprising 28 items, the subscales are categorized into three sections: Functional (F), Ambulation (A), and Instrumental (E).(7) Each activity within the assessment employs a qualitative scale ranging from 0 to 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PHD, Study Chair — Riphah International University
Locations (1):
- Bahawal Victoria Hospital, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No